CLINICAL TRIAL: NCT02826408
Title: A Randomized Placebo Controlled Trial on the Effect of Proton Pump Inhibitors on Palpitations With no Apparent Cause to Explain Such a Symptom
Brief Title: Effect of Proton Pump Inhibitors on Palpitations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Signs and Symptoms
MeSH Terms: conditions — Signs and Symptoms | interventions — Rabeprazole; PACEBO protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active group (Active Comparator): Will receive Rabeprazole sodium (Proton pump inhibitor 20 mg once daily)
  Interventions: Drug: Rabeprazole sodium
- Placebo group (Placebo Comparator): Will receive Folic acid 5 mg once daily
  Interventions: Drug: Pacebo

INTERVENTIONS:
Drug: Rabeprazole sodium — WIll study effect of the medication on palpittions
  Other Names: Active treatment
  Arms: Active group
Drug: Pacebo — Placebo comparison to active treatment
  Arms: Placebo group

SUMMARY:
Palpitation is a common complaint. Patients frequently feel this symptom despite having normal rhythm during symptoms. I have seen many patients who improve significantly on treatment with proton pump inhibitors (PPI). It may be that gastritis provokes a feeling of discomfort that subsequently starts the feeling of palpitation. On searching literature I found no study that investigated the effect of PPI's on palpitations. Therefore I propose a study where the investigators randomize people with palpitations with normal heart rate (no arrhythmia) and no apparent cause such as anxiety or clear illness to receive either PPI or placebo. The result will help to investigate if the improvement is true and if the results are positive this can provide a simple treatment for a common problem.

DETAILED DESCRIPTION:
Methods Two hundred patients with palpitations and no clear cause for their symptoms will be randomized to receive either PPI or placebo for one month. At base line they will be investigated to rule out arrhythmia by documenting normal heart rate (less than 110 beat per minute) or ECG showing normal sinus rhythm or mild sinus tachycardia (Less than 110 per minute) during symptoms. Obvious causes such as anxiety due to a stressful event or organic causes such anemia or thyroid disorders should be also ruled out.

Patient who agree to participate in the study will be asked to sign an informed consent. A baseline questionnaire with symptoms will be filled. They will then be randomized for treatment with either PPI or placebo once at night time. After 10 days of treatment they will be contacted and questioned regarding their symptoms. The two groups will be compared to see if there is any improvement of symptoms with treatment.

Studying group The study will be under the umbrella of the JCC group. Primary investigators are Dr Munir Zaqqa and Dr Ismail Hamam

Support required Pharmaceutical company will be contacted to provide 120 packets with 30 tabs of PPI and if possible packets with similar matching placebo to support the study

Study criteria inclusion

1. Persons with palpitations and no clear cause who are above the age of 16 years and who consent to the study will be included
2. Clear causes that should be excluded are true arrhythmia such SVT or VT or frequent premature atrial or ventricular contractions or any organic cause such as thyroid disorder, anemia (hg less than 11 g/dl) and obvious anxiety disorder
3. Arrhythmia can be excluded by an ECG showing sinus rhythm or sinus tachycardia during episodes or measurement of heart rate by a reliable method during symptoms showing regular heart rate less than 120 beats per minute.
4. Patient will be randomized to either PPI or placebo to be taken one table at night time
5. Patients will be provided with 2 weeks supply but will be evaluated at 10 days to see if symptoms improved
6. The two groups will be compared using statistical methods to see if there is difference in improvement.

Expected harm:

PPI's are generally safe medications. Side effects are rare and generally mild. They include nausea, stomach pain, diarrhea, constipation or headache.

Very rarely allergic reaction can occur with hives, difficulty in breathing and swelling of the face and lips.

Benefit to the patient:

Patients randomized to either group may experience benefit due to the medication or even placebo use. There is no financial benefit of participating in the study. The result of the study will be used to help patient in the future with similar symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Persons with palpitations and no clear cause who are above the age of 16 years and who consent to the study will be included
2. Clear causes that should be excluded are true arrhythmia such SVT or VT or frequent premature atrial or ventricular contractions or any organic cause such as thyroid disorder, anemia (hg less than 11 g/dl) and obvious anxiety disorder
3. Arrhythmia can be excluded by an ECG showing sinus rhythm or sinus tachycardia during episodes or measurement of heart rate by a reliable method during symptoms showing regular heart rate less than 120 beats per minute.
4. Patient will be randomized to either PPI or placebo to be taken one table at night time
5. Patients will be provided with 2 weeks supply but will be evaluated at 10 days to see if symptoms improved
6. The two groups will be compared using statistical methods to see if there is difference in improvement.

Exclusion Criteria:

* Refusal to participate or sign consent form
* Frequency of symptoms less than 2 times per week
* Already taking PPI or H2 blocker

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Palpitations | 2 weeks
  Improvement will be assessed by questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Munir Zaqqa, MD, Principal Investigator — Organizer
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: abstract of study — http://spo.escardio.org/SessionDetails.aspx?eevtid=1220&sessId=21633&subSessId=6401&searchQuery=%2Fdefault.aspx%3Feevtid%3D1220%26days%3D%26topics%3D%26types%3D%26rooms%3D%26freetext%3D%26sort%3D1%26page%3D3%26showResults%3DTrue%26nbPerPage%3D100%26WithWebcast%3D%26WithSlides%3D%26WithAbstract%3D%26WithReport%3D#.WqLNLFRuaDI